CLINICAL TRIAL: NCT02963805
Title: Active City of Liverpool Active Schools and SportsLinx Project: a Clustered Randomised Controlled Trial (The A-CLASS Project)
Brief Title: Active City of Liverpool Active Schools and SportsLinx Project: a Clustered Randomised Controlled Trial
Acronym: A-CLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Teesside University (Other)
Responsible Party: Principal Investigator, Lee Graves, Lecturer, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-SPS-Graves1
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Physical Activity; Health Behavior
Keywords: Children; Physical activity; Physical competence; Obesity; School; Health; Fundamental movement skills
MeSH Terms: conditions — Motor Activity; Health Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- High intensity physical activity (HIPA) (Experimental): Participants attended high intensity vigorous activity after school clubs.
  Interventions: Behavioral: High intensity physical activity (HIPA)
- Fundamental movement skill (FMS) (Experimental): Participants attended fundamental movement skill based after school clubs.
  Interventions: Behavioral: Fundamental movement skill (FMS)
- Physical activity signposting (PASS) (Experimental): Participants attended educational physical activity signposting sessions during school hours.
  Interventions: Behavioral: Physical activity signposting (PASS)
- Control (No Intervention): Children in the control group received British Heart Foundation leaflets that included information on heart health (given to all groups). Children participated in their usual school curriculum including two hours of physical education and school sport per week, both within and beyond the curriculum.

INTERVENTIONS:
Behavioral: High intensity physical activity (HIPA) — This arm consisted of a twice-weekly after-school club at the intervention school for 26 weeks during school term time, delivered by qualified coaches. Each 60 minute session engaged participants in high-intensity vigorous activity using a combination of playground-style games and circuit training activities that aimed to keep children moving and maintain a mean heart rate above 70% of age-predicted maximum heart rate (~145 beats/min) for the session duration. Intensity was verified by heart rate monitoring. Coaches delivered and monitored sessions and increased the intensity over time to allow for the children to progress. The mean heart rate for HIPA sessions was 150 beats/min, with children spending 52 min at this intensity during the session.
  Arms: High intensity physical activity (HIPA)
Behavioral: Fundamental movement skill (FMS) — This arm consisted of a twice-weekly after-school club at the intervention school for 26 weeks during school term time, delivered by qualified coaches. Each 60 minute session focused on improving two skills from the vertical jump, hop, sprint run, dodge, kick, catch, overarm throw, and strike. All skills were taught in equal quantities. Each session was designed to maximise participation and enjoyment, and consisted of various games, drills, self-learning activities, and offered numerous opportunities for practice. Skill components were taught to the children using simple learning cues, and skill related questions were used to develop purposeful feedback. The mean heart rate for FMS sessions was recorded at 141 beats/min, with children spending 55 min at this intensity during the session.
  Arms: Fundamental movement skill (FMS)
Behavioral: Physical activity signposting (PASS) — A researcher visited participants once per week in 6 weekly blocks to set an activity mission to complete outside school with family and friends. Twenty missions were set over 4 x 6 week blocks, each separated by a 6 week break. Each mission suggests a task as a prompt to participate in physical activity and decrease sedentariness during the week. Children received a sticker on a wall chart for returning the mission; children were rewarded with prizes if all missions were returned in each block. If all missions were returned in a block, a reward was given. 58% of children returned all twenty missions. In addition to the missions, pedometers were issued as a promotional tool for the duration of the project for self-monitoring of activity.
  Arms: Physical activity signposting (PASS)

SUMMARY:
The purpose of the A-CLASS project was to measure the effect of the 4 hour offer on children's physical activity, health and physical competence.

DETAILED DESCRIPTION:
Study design

Treatment arms in this four-arm parallel-group cluster randomised controlled trial (RCT) included a high intensity physical activity (HIPA) intervention group, a fundamental movement skill (FMS) intervention group, a physical activity signposting (PASS) intervention group and a control group (usual practice).

Recruitment

- Organisation level

Sixteen primary schools were targeted by the research team in May-July 2006. The schools were targeted based on their size (student enrolment >400 primary school; >250 junior school), current afterschool club provision (limited), school sport facilities available for use (bi-weekly) and socioeconomic status of the school postcode classified by postcode in the Index of Multiple Deprivation as deprived (IMD > 40). Signed consent was sought and obtained from the head teachers of the sixteen schools for pupil recruitment, study contact, laboratory visits during school time and access to school facilities. Eight from the sixteen schools were randomly selected to take part using random number allocation.

- Individual level

All children in year 5 in consenting schools received a verbal and written overview of the study through a researcher led study information session held at the respective schools. Children were given 2 weeks to express interest via the return of a written assent form (children) and parental/guardian consent form to their school teacher. Medical questionnaires were distributed to all children who agreed to take part in the study, and they were assessed for stature and body mass in order to calculate body mass index (BMI; kg/m2). BMI was used as guide to target the children who were overweight or may be nearing overweight according to BMI cut-off thresholds stipulated by Chinn and Rona (2004). Generally, 20-25 children with the highest BMI within each school who were free from the presence of chronic disease, metabolic disorders, motor or co-ordination difficulties and prescribed medications including steroids inhaled by asthma sufferers were then enrolled to participate in the project. There was no racial or gender bias in the selection of participants.

Group assignment and Intervention

Participating schools were randomly allocated by a computer generated procedure to one of four treatments to reduce risk of contamination effects across the trial.

Data collection

Measurements took place at three time points: at baseline (month 0; September to mid-October 2006); end-intervention (9 months; June to mid-July 2007); and follow-up (3 years; October 2009). At each time point participants attended University laboratories for individual assessments. At each time point participants' habitual physical activity was objectively assessed using accelerometers, and participants' fundamental movement skills were assessed at their respective school. Prior to laboratory visits, participants were instructed to fast for a minimum of 8 hours and avoid strenuous exercise for 24 hours.

Sample size

It was feasible to recruit eight schools and randomly assign two schools to each of the four arms. With an estimated number of consenting Year 5 pupils of 20 per school, the planned sample size was around 40 participants per arm. Allowing for 10% attrition at 9 months and a design effect of 1.2 to account for school-level clustering (ICC of 0.01), our effective sample size was 30 participants per arm. This sample size provides approximately 80% power at 2P=0.05 to detect a targeted difference between intervention and control (3 planned comparisons) at the 9-month timepoint of 3 units for the total FMS skills score (based on an between-subjects standard deviations (SD) of 7 units and a reliability of r=0.8 over the timeframe of the intervention; ANCOVA model adjusting for baseline FMS score). With an anticipated attrition of up to 50% for the 2-year follow-up timepoint, our effective sample size was only 16 participants per arm. Group comparisons at this timepoint are therefore defined as exploratory, as we have relatively low power to detect the same effect size (around 50%).

Statistical analyses

There are too few clusters per arm to account robustly for the hierarchical data structure using linear mixed (multilevel) modelling, generalised estimating equations, or clustered robust standard errors. Therefore, data will be analysed at the individual level, with standard errors inflated by the square root of the design effect. The change in FMS score from baseline to post-intervention (9-months) will be compared between arms using a regression model (ANCOVA), adjusting for baseline FMS score and sex. There are 3 planned comparisons comprising each of the 3 interventions vs. usual practice. Point estimates will be derived together with uncertainty expressed as 90% confidence intervals. For the primary outcome, a purely exploratory sub-group analysis will be conducted using a sex-by-intervention group interaction term to examine the potential for differential intervention effects in boys vs. girls. Secondary outcomes will be analysed using the same general modelling approach, but with no inferential emphasis placed on the results. Where appropriate, a principled method will be applied to address missing data (e.g., multiple imputation or full information maximum likelihood).

ELIGIBILITY:
Inclusion Criteria:

a. body mass index (BMI) score within the lower 50th percentile relative to children in their year at their school.

Exclusion Criteria:

1. family history of sudden death.
2. presence of chronic disease, metabolic disorders, motor or co-ordination difficulties
3. prescribed medications including steroids inhaled by asthma sufferers

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total skills score at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  8 fundamental movement skills were assessed (vertical jump, sprint run, hop, dodge (locomotor) kick, catch, overarm throw, strike (object-control). Assessments were conducted in the school playground or gym (weather dependent) by one researcher with the same equipment at each site. Children were given a verbal description and single demonstration of the skill. Children performed each skill 5 times (3 for the sprint run and dodge) in a standardised order. Recordings of all participants were taken from identical angles and distances using a tripod mounted video camera.
  Skills were assessed by video analysis using process-orientated measures. If the skill component was present on 4 out of 5 trials (2 out of 3 for sprint run and dodge) the child was marked as possessing that skill component. The number of skill components checked as present in each of the 8 skills was summed to create an overall skill score (max score 48) for use in the analysis.

SECONDARY OUTCOMES:
Change from baseline in body mass index at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Calculated from assessment of stature and body mass
Change from baseline in bone mineral content of the total body at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in bone areal density of the total body at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in bone mineral content of the femoral neck at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in bone areal density of the femoral neck at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in bone mineral content of the lumbar spine at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in bone areal density of the lumbar spine at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in fat mass at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in lean tissue mass at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in percentage body fat at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in visceral fat at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via dual-energy x-ray absorptiometry
Change from baseline in triceps skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in subscapular skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in biceps skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in iliac crest skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in supraspinale skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in abdomen skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in front thigh skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in medial calf skinfold thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in waist circumference at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in gluteal circumference at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in arm girth relaxed at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in arm girth flexed and tensed at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in calf girth at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in bone breadth on the biepicondyles of the humerus at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in bone breadth on the biepicondyles of the femur at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard International Society for the Advancement of Kinanthropometry (ISAK) techniques
Change from baseline in proficiency of the vertical jump at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the sprint run at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the hop at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the dodge at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the kick at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the catch at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the overarm throw at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in proficiency of the strike at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via video analysis
Change from baseline in systolic blood pressure at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via an automated sphygmomanometer
Change from baseline in diastolic blood pressure at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via an automated sphygmomanometer
Change from baseline in left ventricular structures at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via echocardiography
Change from baseline in left ventricular mass at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via echocardiography
Change from baseline in carotid artery intima media thickness at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via standard ultrasound techniques
Change from baseline in peak oxygen uptake at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via discontinuous incremental treadmill protocol to volitional exhaustion
Change from baseline in sedentary time at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via accelerometry
Change from baseline in light intensity physical activity at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via accelerometry
Change from baseline in moderate intensity physical activity at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via accelerometry
Change from baseline in vigorous intensity physical activity at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via accelerometry
Change from baseline in steps taken at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via accelerometry
Change from baseline in physical self perceptions at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via the Children and Youth Physical Self-Perception Profile (CY-PSPP)
Change from baseline in perceived competence in fundamental movement skills at end intervention (9 months) and follow up (3 years) | Baseline (month 0), End-intervention (9 months), Follow-up (3 years)
  Assessed via an adapted questionnaire from a previous trial

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Stratton, PhD, Study Chair — Swansea University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McWhannell N, Foweather L, Graves LEF, Henaghan JL, Ridgers ND, Stratton G. From Surveillance to Intervention: Overview and Baseline Findings for the Active City of Liverpool Active Schools and SportsLinx (A-CLASS) Project. Int J Environ Res Public Health. 2018 Mar 23;15(4):582. doi: 10.3390/ijerph15040582. PMID 30720781